CLINICAL TRIAL: NCT04049123
Title: A Study to Evaluate the Pharmacokinetics and Glucodynamics of LY900014 Following Single Dose Administration in Healthy Chinese Subjects
Brief Title: A Study of LY900014 in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16644; I8B-MC-ITRY (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Healthy
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Insulin Lispro (Humalog) (Active Comparator): 15 units (U) Insulin Lispro (Humalog) administered once, subcutaneously (SC), in one of three study periods.
  Interventions: Drug: Insulin Lispro
- LY900014 (Experimental): 7 U, and 15 U LY900014 administered once, SC, in two of three study periods.
  Interventions: Drug: LY900014

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014
Drug: Insulin Lispro — Administered SC
  Other Names: LY275585; Humalog
  Arms: Insulin Lispro (Humalog)

SUMMARY:
The purpose of this study is to evaluate a new formulation of insulin lispro, LY900014, which is a drug that lowers blood sugar. The study will look at how the body processes LY900014 and the effect of LY900014 on blood sugar levels. For each participant, the study will consist of 3 periods and will last about 51 days.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy native Chinese males or females
* Female participants:

  * Women of child-bearing potential who are abstinent or use effective methods of contraception for the entirety of the study.
  * Women not of child-bearing potential who are infertile or post-menopausal
* Have a body mass index (BMI) of 18 to 28 kilograms per square meter (kg/m²)
* Are nonsmokers
* Have a fasting plasma glucose value >71 milligrams per deciliter (mg/dL) (3.9 millimoles per liter [mmol/L]) and <108 mg/dL (6.0 mmol/L)

Exclusion Criteria:

* Are currently enrolled in a clinical study, or have participated, within the last 30 days, in a clinical study involving an investigational product
* Have previously completed or withdrawn from this study or any other study investigating LY900014
* Have known allergies to LY900014 or any components of the formulation
* Have a significant history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data
* Intend to use over-the-counter or prescription medication within 7 and 14 days, respectively, prior to dosing or during the study.
* Have donated blood of more than 400 milliliters (mL) within the previous 6 months of study screening or donated more than 100 mL within the last 30 days.
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- West China Hospital Sichuan University, Chengdu, Cn-51, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 3-period crossover study in which participants received a single 7 Unit (U), and a single 15 U subcutaneous (SC) dose of LY900014 in two of three dosing sequences, and 15 U SC dose of Humalog in one of three dosing sequences. There was a washout period of ≥ 3 days between euglycemic clamp visits.
Groups:
- Sequence 1: CAB: Participants received a single SC dose in each treatment period.
  C = 15 U Humalog
  A = 7 U LY900014
  B = 15 U LY900014
- Sequence 2: ACB: Participants received a single SC dose in each treatment period.
  A = 7 U LY900014
  C = 15 U Humalog
  B = 15 U LY900014
- Sequence 3: ABC: Participants received a single SC dose in each treatment period.
  A = 7 U LY900014
  B = 15 U LY900014
  C = 15 U Humalog
Period: Period 1
Arm/Group | Sequence 1: CAB | Sequence 2: ACB | Sequence 3: ABC
Started | 5 | 5 | 5
Received at Least One Dose of Study Drug | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1: CAB | Sequence 2: ACB | Sequence 3: ABC
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1: CAB | Sequence 2: ACB | Sequence 3: ABC
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants whether or not they completed all protocol requirements.
Groups:
- Overall Baseline: Participants received a single 7 U, and a single 15 U SC dose of LY900014 in 2 of 3 periods and 15 U SC dose of Humalog in 1 of 3 periods.
Arm/Group | Overall Baseline
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 15

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Serum Concentration Versus Time Curve From Time Zero to 10 Hours Postdose (AUC[0-10h])
Description: PK: Insulin Lispro AUC(0-10h)
Time Frame: Day 1: Predose, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, 60, 70, 90, 120, 150, 180, 240, 300, 360, 420, 480, 540, and 600 minutes postdose
Population: All participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole * hour per Liter (pmol*h/L)
Groups:
- 7 U LY900014: Single SC dose 7 U LY900014.
- 15 U LY900014: Single SC dose 15 U LY900014.
- 15 U Humalog: Single SC dose 15 U Humalog.
Arm/Group | 7 U LY900014 | 15 U LY900014 | 15 U Humalog
Number analyzed (Participants) | 15 | 15 | 15
picomole * hour per Liter (pmol*h/L) | 708 (12) | 1580 (11) | 1600 (12)

2. Secondary Outcome: Pharmacodynamics (PD): Total Amount of Glucose Infused (Gtot)
Description: Gtot is the total amount of glucose infused over the duration of the clamp procedure (10 hours) for each study period.
Time Frame: Day 1: Predose: -10, -20, -30 minutes; During clamp: every 2.5 to 3 minutes for the first 30 minutes; every 5 minutes for 30 to 120 minutes; every 10 minutes for 120 to 480 minutes and every 20 minutes for 480 to 600 minutes postdose
Population: All participants who received at least one dose of study drug and had evaluable glucodynamic (GD) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram per kilogram (mg/kg)
Arm/Group | 7 U LY900014 | 15 U LY900014 | 15 U Humalog
Number analyzed (Participants) | 15 | 15 | 15
milligram per kilogram (mg/kg) | 989 (35) | 1540 (40) | 1720 (32)

ADVERSE EVENTS:
Time Frame: Baseline to end of study (up to 183 days).
Description: All enrolled participants, whether or not they completed all protocol requirements.
Groups:
- 7 Unit (U) LY900014: Single subcutaneous (SC) dose 7 U LY900014.
Arm/Group | 7 Unit (U) LY900014 | 15 U LY900014 | 15 U Humalog
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 4/15 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 7 Unit (U) LY900014 (N=15) | 15 U LY900014 (N=15) | 15 U Humalog (N=15)
Nodal rhythm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT04049123/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT04049123/SAP_001.pdf